CLINICAL TRIAL: NCT07187700
Title: Developing Trustworthy Artificial Intelligence (AI)-Driven Tools to Predict Vascular Disease Risk and Progression: the Prospective VASCUL-AID Study
Acronym: VASCUL-AID-PRO
Status: Not yet recruiting | Type: Observational
Sponsor: Amsterdam UMC (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Brightfish (Unknown); Technical University of Twente (Other); Universidade do Porto (Other); Aveiro University (Other); Centro Hospitalar De São João, E.P.E. (Other); Stichting Allai (Unknown); University of Belgrade (Other); Hospital District of Helsinki and Uusimaa (Other); VINČA INSTITUTE OF NUCLEAR SCIENCES Belgrado (Unknown); University of Bergen (Other); Asklepios Kliniken Hamburg GmbH (Other); Centre Hospitalier Universitaire de Nice (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Associate Prof. Dr. Kak Khee Yeung, Prof. Dr., Amsterdam UMC
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: 2025.0042
Record Dates: First submitted 2025-08-13; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Abdominal Aorta Aneurism; Peripheral Arterial Disease
Keywords: Abdominal aortic aneurysm; peripheral arterial disease; artificial intelligence; cardiovascular risk; prediction models; disease progression
MeSH Terms: conditions — Peripheral Arterial Disease; Aortic Aneurysm, Abdominal; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Whole blood, blood plasma, aorta tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AAA: * Males/females between 40 and 90 years of age.
  * Males and females with AAA at inclusion, any diameter >3 cm (or 1.5x larger than their non-dilated part of the aorta).
  * Include: infrarenal, juxtarenal, pararenal, suprarenal abdominal aortic aneurysms.
  Without prior AAA surgery or or planned AAA surgery within 6 months after inclusion.
- PAD: * Males/females between 40 and 90 years of age.
  * Patients with peripheral arterial disease stage Fontaine 2a and 2b at inclusion. Medical history (e.g. CLTI) does not matter, current disease stage is leading at inclusion.

SUMMARY:
Introduction:

Peripheral arterial disease (PAD) and abdominal aortic aneurysm (AAA) are vascular conditions associated with significant morbidity and mortality, with 25% of AAA patients and 23% of PAD patients being at a high risk of developing cardiovascular disease. Cardiovascular risk management can reduce the risk of major adverse cardiovascular events in AAA patients from 43% to 14%. However, cardiovascular risk is not always adequately addressed in these patients. The VASCUL-AID-PRO study aims to deliver clinically relevant prediction models using artificial intelligence and machine learning of patient outcomes to enable personalized management of vascular disease.

Method:

VASCUL-AID-PRO is a multi-centre international prospective cross-sectional study aiming to include 500 AAA patients and 600 PAD patients across 6 European centres. The aim is to achieve a follow-up time up to 4 years.

The study will include individuals aged 40-90 with either an abdominal aortic aneurysm (infrarenal, juxtarenal, pararenal, or suprarenal abdominal aortic aneurysm) or Fontaine stage 2 peripheral arterial disease.

The VASCUL-AID-PRO study will gather a variety of data from all participants, including clinical data, blood and tissue samples, cardiovascular lab values, imaging data, electrocardiograms, data from wearables and quality of life.

This data gathered will be used to further develop the multi model prediction models being developed on 5000 AAA and 6000 PAD patients included in the currently ongoing VASCUL-AID-RETRO study, with the aim of providing a clinically relevant prediction models of disease progression and other cardiovascular disease for AAA and PAD patients.

Furthermore, the models developed in the VASCUL-AID studies will be internally validated using a subset of patients from the VASCUL-AID-PRO study.

Ethical considerations:

Ethical and legal considerations are paramount throughout the VASCUL-AID project. To address these concerns, an ELSI framework will be developed and integrated into all stages of the project. This framework will be continuously updated to ensure alignment with evolving ethical, legal, and social standards. This framework will specifically focus on patient safety, data handling, AI regulation and implementation, and potential biases associated with AI.

ELIGIBILITY:
Inclusion Criteria AAA:

* Males/females between 40 and 90 years of age.
* Males and females with AAA at inclusion, any diameter >3 cm (or 1.5x larger than their non-dilated part of the aorta).
* Include: infrarenal, juxtarenal, pararenal, suprarenal abdominal aortic aneurysms.

Exclusion Criteria AAA:

Patients with:

* Insufficient schooling or sensorial deficits that interfere understanding informed consent.
* Not able to use the VASCUL-AID mobile health app (that will be provided in Dutch, English, German, Portuguese, Serbian, Finish, Swedish languages).
* Proven or highly suspected for infected, mycotic AAA
* Previous AAA surgery or planned for an AAA surgery within 6 months
* Ruptured AAA

Inclusion Criteria PAD:

* Males/females between 40 and 90 years of age.
* Patients with peripheral arterial disease stage Fontaine 2a and 2b at inclusion. Medical history (e.g. CLTI) does not matter, current disease stage is leading at inclusion.

Exclusion Criteria PAD:

Patients with:

* Insufficient schooling or sensorial deficits that interfere understanding informed consent.
* Not able to use the VASCUL-AID mobile health app (provided in Dutch, English, German, Portuguese, Serbian, Finnish, Swedish languages).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 AAA patients and 100 PAD will be included per clinical center, with exeption for Asklepios Hamburg, they will solely include 100 PAD patients.
  This comes to a total of 1100 patients across 6 clinical centers in Europe.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Development and internal validation of AI-driven tools to predict high or low risk disease progression in AAA and PAD. | From baseline to 4 years follow-up.
  The VASCUL-AID AI tools aim to predict AAA (rupture, mortality, cerebrovascular accident) and PAD (mortality, myocardial infarction, major amputation) progression, MACE and MALE.
  The internal validation is done by comparing the predicted disease progression, MACE, MALE and mortality rates with actual disease progression.

SECONDARY OUTCOMES:
Accuracy of developed VASCUL-AID driven algorithms that classify AAA patients according to high or low risk disease progression. | From baseline to 4 years follow-up
  Accuracy of developed VASCUL-AID AI-driven algorithms that classify AAA patients according to high or low risk disease progression and MACE. In addition, models will be developed on the other predefined outcomes from the core outcome set, these include: clinical success after an operation [yes/no], graft infection after an operation [yes/no], reintervention [yes/no], the AAA can be treated through endovascular treatment [yes/no], adherence to prescribed drugs [yes/no], secondary prevention, treatment options and complications.
Accuracy of developed VASCUL-AID driven algorithms that classify PAD patients according to high or low risk disease progression. | From baseline to 4 years follow-up
  Accuracy of developed VASCUL-AID AI-driven algorithms that classify PAD patients according to high or low risk disease progression, MALE and MACE. In addition, models will be developed on the other predefined outcomes from the core outcome set, these include: acute limb ischemia [yes/no], thromboembolic complications [yes/no], disease progression [yes/no], pain-free walking distance [meters], physical activity, smoking cessation, secondary prevention, treatment options and complications.
Patient reported outcome measures for AAA and PAD. | From baseline to 4 years follow-up.
  Good communication by healthcare worker about diagnosis [Questionnaires].
Patient reported outcome measures for health-related quality of life. | From baseline to 4 year follow-up.
  Numeric (Pain) Rating Scale (0-10, no pain to most intense pain).
Patient reported outcome measures for health-related quality of life. | From baseline to 4 year follow-up
  PROMIS Scale v1.2 - Global Health measure. Answer rank on a scale of 0-5, with the higher score being more preferred.
Patient reported outcome measures for health-related quality of life. | From baseline to 4 years follow-up.
  EQ-5D-5L Euroqol questionnaire.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Patient reported outcome measures for vascular quality of life for PAD. | From baseline to 4 year follow-up
  Vascular Quality of Life Questionnaire (VascuQol) consists of 25 questions regarding the QoL in patients with vascular diseases, regarding activity level, symptoms, pain, emotion and social consequences. It uses a 7-point Likert scale, where a low score equels a severe sense of limitations.
Patient reported outcome measures for AAA related quality of life. | From baseline to 4 year follow-up.
  AneurysmDQoL - Abdominal Aortic Aneurysm Quality of Life
  The AneurysmDQoL is a 24-item measure including two overview items designed for audit purposes which measure generic 'present QoL' and AAA-specific 'impact of AAA on QoL'. A further 22 items measure the impact of having an abdominal aortic aneurysm on specific aspects of life and the importance of these aspects of life for QoL. In addition the questionnaire includes a free-text item. This allows patients to comment on any other QoL domains not covered in the questionnaire.
Questions regarding medical status. | From baseline to 4 year follow-up
  A custom list of questions developed to gather all changes in medical history of the patients.
6-minute walking test questionnaire | From baseline to 4 year follow-up
  The 6-minute walking test is a test in which patients are asked to walk for a duration of 6 minutes and then report the distance they have walked in that time and whether they experienced any complaints.
Medication use questionnaire | From baseline to 4 year follow-up
  Asks the patient to write down all active medication.
Smoking cessation questionnaire | From baseline to 4 year follow-up.
  A custom list of questions asking patients about smoking cessation and how they are managing quitting.
Questionnaire regarding health-care provider communication. | From baseline to 4 year follow-up.
  This questionnaire scores how well the patient experienced contact with their health care provider. Each question is answered on a scale between strongly agree - strongly disagree.
Cost-effectiveness and Clinical Implementation Study | baseline to 4 years follow-up
  The project will include data collection of costs and Health-Related Quality of Life (HRQoL) prospectively. The economic analysis will be performed in accordance with the Consolidated Health Economic Evaluation Reporting Standards (CHEERS) statement. An estimation of costs and HRQoL progression until MACE will be performed and descriptive statistics will be used to describe their respective evolution (up to 4 years).
  To describe the evolution and further estimate threshold where the implementation of VASCULAID within hospitals could be more efficient, the number of patients with at least one MACE during the follow-up period will be used to estimate the costs and HRQoL per event among the dedicated subgroup of population where HRQoL is collected. Only direct costs will be considered in the analysis.
  The result will be expressed in euros per patient (then distinguishing MACE vs free of MACE) over the follow-up. QALYs will be expressed per patients.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. K.K. Yeung, MD, PhdD, FEBVS, Principal Investigator — Amsterdam UMC

IPD SHARING:
Plan to Share IPD: Yes
Patient data will be pseudoanonymised and recorded in an eCRF provided in the web-based app, a secured central data system conform EU GDPR guidelines hosted by Brightfish B.V. (certified: ISO 27001, NEN751-012, ISC121, ISO9001:2015; QSC808).
  The collected data consists of heart-rate data, blood pressure values, clinical questionnares, medical records, medical imaging, blood samples for proteomics, lipidomics and genomics analyses results, demographics.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data sharing agreement was signed by all parties in August 2024 and shall remain in force for the period of the Project, unless terminated earlier
Access Criteria: All partners in the VASCUL-AID consortium through the Brightfish system and through XNAT for medical imaging.

REFERENCES:
- See also: The consortium website with further information regarding the incorporated studies. — https://vascul-aid.eu/